CLINICAL TRIAL: NCT03720171
Title: An Osseointegrated Transfemoral Prosthesis Study Evaluating Stable Neural Signal Transmission in Patients With Transfemoral Amputations
Brief Title: e-OPRA Implant System for Lower Limb Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrum (Industry)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDE G170304
Record Dates: First submitted 2018-10-19; First posted 2018-10-25 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Amputation
Keywords: Osseointegration; Bone-anchored prosthesis; Neuro-prosthesis

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, uncontrolled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- e-OPRA Implant System (Experimental): Implantation of e-OPRA Implant System in lower limb.
  Interventions: Device: e-OPRA Implant System

INTERVENTIONS:
Device: e-OPRA Implant System — Implantation of e-OPRA Implant System in lower limb to be used with amputation limb prosthesis

SUMMARY:
The e-OPRA Implant System, is a further development of the OPRA (Osseointegrated Prostheses for the Rehabilitation of Amputees) Implant System, approved under HDE (Humanitarian Device Exemption) H080004. The e-OPRA Implant system is an implant system for direct skeletal anchorage of amputation prostheses. The added feature in the e-OPRA Implant system, is a bidirectional interface into the human body that allows permanent and reliable communication using implanted electrodes. These electrodes will provide long-term stable bioelectric signals for an improved control of the prosthetic limb. The purpose of the study is to evaluate the feasibility of a lower limb amputee with the e-OPRA Implant System exhibiting full neural control over a neuro-mechanical prosthetic system.

A maximum of six subjects will be enrolled. Each subject will undergo a surgery where the e-OPRA Implant System will be implanted. The subjects will participate in follow-up sessions of which the last one occurs approximately 24 months after the surgery. This is a prospective, non-randomized, uncontrolled study.

ELIGIBILITY:
Inclusion Criteria:

A potential subject will be included in the study if she/he meets all of the following inclusion criteria:

* Male or Female age 22-65 at the time of surgery.
* The patient must have a medical condition requiring performance of a unilateral transfemoral amputation with a minimum of 13 cm of residual femur after amputation, and:

A: At a minimum level of amputation of 20 cm or greater above the knee joint line if physical therapy and prosthetist evaluation is commensurate with a standard K3 ambulatory status; or, B: At a minimum level of amputation of 16 cm above the knee joint line as part of a single-stage procedure if physical therapy and prosthetist evaluation is commensurate with a more active K3 or less active K4 postoperative ambulatory status.

* The subject must have undergone independent consultation with at least two lower extremity surgical specialists to ensure they have exhausted all limb salvage options prior to undergoing amputation, as well as a psychiatric evaluation to ensure appropriate capacity and volition.
* The patient must have the ability to ambulate at variable cadence (an expected lower extremity prosthesis functional level of K3 or above).
* The patient must have adequate bone stock to support the implanted device.
* In the opinion of the investigators, normal cognitive function and absence of any physical limitations, addictive diseases or underlying medical conditions that may preclude patient from being a good surgical and/or study candidate.
* Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study including the prescribed rehabilitation program.
* Written informed consent to participate in the study provided by the patient or legal representative.

Exclusion Criteria:

* Women who are pregnant, lactating or planning a pregnancy during the first twelve (12) months of the post-surgical follow-up.
* Subjects who have not been completely abstinent from tobacco use for at least 6 weeks preoperatively.
* Active infection or dormant bacteria.
* Subjects would have less than 2 mm of remaining cortex bone available around the implant, if implanted.
* Evidence of or a documented history of severe peripheral vascular disease, diabetes mellitus (type I or type II), skin diseases, Neuropathy or neuropathic disease and severe phantom pain, or osteoporosis, such that, in the opinion of the investigator, will not allow the subject to be a good study candidate.
* Evidence of any active skin disease involving the proposed surgical limb.
* History of systemically administered corticosteroids, immune-suppressive therapy or chemotherapy drugs within six (6) months of implant surgery.
* Severe co morbidity, atypical skeletal anatomy, or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, shortened life expectancy, vulnerable patient population, BMI >40, etc.).
* The patient is currently involved in another clinical study where that participation may conflict or interfere with the treatment, follow-up or results of this clinical study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-03-08 (Actual)

PRIMARY OUTCOMES:
Electrode function | 24 months
  i) To evaluate implantation robustness, and connector/lead integrity:
  i.a. Measured Impedance (kOhms)
  i.b. Maximal Voluntary Contraction (MVC) Amplitude (mV)
  ii) To evaluate sensor function and signal quality:
  ii.a. Signal-to-noise ratio (SNR) above 2

SECONDARY OUTCOMES:
Preferred walking speed | 24 months
  Preferred walking speed, as each subject ambulates with the neuromechanical prosthesis, will be evaluated. Preferred walking speed will be compared to a non-amputee height/weight match for each enrolled subject. A baseline data set will first be collected for each subject ambulating with a conventional prosthesis. Each subject will be timed as they traverse a predetermined distance at a steady speed that they deem most comfortable.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh M Herr, PhD, Principal Investigator — Massachusetts Insititute of Technology
Locations (1):
- MIT Media Lab, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No